CLINICAL TRIAL: NCT07277478
Title: Effects of Auricular Acupressure on Relieving Pain in Postpartum Women With Episiotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HSIAO AI WEN (Other)
Responsible Party: Sponsor-Investigator, HSIAO AI WEN, Nurse, Fu Jen Catholic University Hospital
Organization: Fu Jen Catholic University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FJUH113431
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Auricular Acupressure; Episiotomy Pain
Keywords: episiotomy; auricular acupressure; pain; impact on daily life; satisfaction with pain management
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: participants were postpartum women who had undergone episiotomy and were randomly assigned to the intervention or control group using an Excel-generated random allocation table. A total of 90 patients were enrolled, with 4 excluded, resulting in 43 participants in each group. Demographic data were collected before the intervention. After placental delivery, the intervention group received routine care plus a transparent patented auricular patch containing magnetic beads, while the control group received a transparent patented auricular patch without magnetic beads. The selected acupoints included internal genitalia (TF2), external genitalia (HX4), Shenmen (TF4), sympathetic (AH6a), and subcortex (AT4).
Who Masked: Participant
Masking Description: This study design was a randomized controlled single-blind trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- auricular patch containing magnetic beads (Experimental): After placental delivery, the intervention group received routine care plus a transparent patented auricular patch containing magnetic beads, while the control group received a transparent patented auricular patch without magnetic beads. The selected acupoints included internal genitalia (TF2), external genitalia (HX4), Shenmen (TF4), sympathetic (AH6a), and subcortex (AT4).
  Interventions: Device: auricular patch
- auricular patch without magnetic beads (Placebo Comparator): After placental delivery, the intervention group received routine care plus a transparent patented auricular patch containing magnetic beads, while the control group received a transparent patented auricular patch without magnetic beads. The selected acupoints included internal genitalia (TF2), external genitalia (HX4), Shenmen (TF4), sympathetic (AH6a), and subcortex (AT4).
  Interventions: Device: auricular patch

INTERVENTIONS:
Device: auricular patch — After placental delivery, the intervention group received routine care plus a transparent patented auricular patch containing magnetic beads, while the control group received a transparent patented auricular patch without magnetic beads. The selected acupoints included internal genitalia (TF2), external genitalia (HX4), Shenmen (TF4), sympathetic (AH6a), and subcortex (AT4)

SUMMARY:
This randomized, single-blind controlled trial examined the effects of auricular acupressure on postpartum women who underwent episiotomy. A total of 86 participants were allocated to either an intervention group, which received routine care plus transparent auricular patches containing magnetic beads applied to selected acupoints, or a control group, which received identical patches without magnetic beads. The patches were applied for 48 hours after delivery. Perineal pain and its impact on daily activities were assessed at 2, 12, 24, and 48 hours postpartum, while satisfaction with perineal pain care was measured at 48 hours. Using independent t-tests, chi-square tests, and generalized estimating equations, the study evaluated whether auricular acupressure reduced perineal wound pain, lessened pain-related interference with daily activities, and improved satisfaction with perineal pain management.

ELIGIBILITY:
-Inclusion Criteria-

1. Women with singleton pregnancies who delivered vaginally.
2. Women who underwent episiotomy.
3. Gestational age between 37 and 42 weeks.
4. Willing to participate in the study and provide signed informed consent.
5. Age 18 years or older.

-Exclusion Criteria-

1. Women with skin lesions or allergies at the auricular acupressure site.
2. Women with gynecological disorders, such as uterine fibroids, adenomyosis, or endometriosis.
3. Women or newborns with severe postpartum complications, such as postpartum hemorrhage, infection, perineal hematoma, major neonatal diseases, or admission to the neonatal intensive care unit.
4. Women with psychiatric disorders, such as anxiety or depression.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-12-07 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
perineal pain | At 2, 12, 24, and 48 hours postpartum
  Structured questionnaires were used to assess perineal pain and its impact on daily activities at 2, 12, 24, and 48 hours postpartum.

SECONDARY OUTCOMES:
impact on daily life | At 2, 12, 24, and 48 hours postpartum
  Structured questionnaires were used to assess perineal pain and its impact on daily activities at 2, 12, 24, and 48 hours postpartum.
satisfaction with pain management | At 48 hours postpartum
  At 48 hours postpartum, and satisfaction with perineal pain care at 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: AI WEN HSIAO, Study Chair — National Taipei University of Nursing and Health Sciences
Locations (1):
- Hsiao Ai Wen, Taipei, Sanchong, Taiwan

IPD SHARING:
Plan to Share IPD: No